CLINICAL TRIAL: NCT01758302
Title: A Pilot Laboratory Study Investigating How Physical Tasks and Hunger Affect Taste Perception
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2T32HL076134-06XX; 2T32HL076134-06 (NIH)
Record Dates: First submitted 2012-12-19; First posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-12

CONDITIONS: Food Consumption; Perseverance
Keywords: taste test; food consumption; hunger
MeSH Terms: interventions — Vegetables

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- No physical task + Taste cookies (Active Comparator): Participants in this arm do not engage in a physical activity task. They are asked to taste test chocolate chip cookies.
  Interventions: Other: Cookies; Behavioral: No physical task
- No physical task + Taste vegetable (Active Comparator): Participant does not complete a physical activity. Asked to taste test raw celery or radishes.
  Interventions: Other: Vegetables; Behavioral: No physical task
- Simple physical task + Taste vegetables (Active Comparator): Participants are asked to complete a simple physical task and are asked to taste test raw celery or radishes.
  Interventions: Behavioral: Simple physical task; Other: Vegetables
- Complex physical task + Taste vegetables (Active Comparator): Participants complete a more complex physical task that is novel and challenging. They are asked to taste test raw celery or radishes.
  Interventions: Behavioral: Complex physical task; Other: Vegetables

INTERVENTIONS:
Behavioral: Simple physical task — Participants are asked to complete a 1-time simple physical task that is not challenging nor novel (moving small objects across a room).
  Arms: Simple physical task + Taste vegetables
Behavioral: Complex physical task — Participants are asked to complete a 1-time physical task that is low intensity but somewhat complex (involves a novel request to move objects in a way that is challenging and requires some coordination).
  Arms: Complex physical task + Taste vegetables
Other: Cookies — Participants are asked to taste test chocolate chip cookies
  Arms: No physical task + Taste cookies
Other: Vegetables — Participants are asked to taste test raw celery or radishes
  Arms: Complex physical task + Taste vegetables; No physical task + Taste vegetable; Simple physical task + Taste vegetables
Behavioral: No physical task — As a control, for 2 of the arms, participants are not asked to engage in a physical task
  Arms: No physical task + Taste cookies; No physical task + Taste vegetable

SUMMARY:
This one time pilot laboratory study focuses on examining the relationship between different types of physical tasks and taste perception of high and low-calorie foods among hungry individuals.

ELIGIBILITY:
Inclusion Criteria:

* Willing to travel to laboratory around lunchtime for the study
* Willing to abstain from eating and drinking caloric beverages for at least 4 hours prior to completing the study
* Typically eats lunch

Exclusion Criteria:

* Diabetes, eating disorder, or any other condition that makes it unadvisable for participant to refrain from eating or drinking caloric beverages for 4 hours.
* Food allergies that would prevent participants from eating chocolate chip cookies or vegetables
* Pregnant or lactating
* Typically goes for longer than 5 hours (not counting sleep time) between meals and snacks
* Physical disabilities that would make it difficult for the participant to walk or to use their hands to grasp objects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
physical perseverance | 1 hour
  as measured via maintained grip using a hand dynamometer on the dominant hand and set to 70% of participant's maximum grip strength

SECONDARY OUTCOMES:
food preference | 1 hour
  Food preference measured via participant's reported ratings after tasting different food.
Amount of food eaten | 1 hour
  Amount of food that participants eat will be measured via a food scale at the end of the study.
Mood | 1 hour
  Participant's subjective mood will be measured using a mood questionnaire (PANAS).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomeng Xu, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States